CLINICAL TRIAL: NCT00992524
Title: Oral Misoprostol Titrated Solution Versus Vaginal Misoprostol for Induction of Labour: Randomized Controlled Trial
Brief Title: Oral Titrated Misoprostol for Induction of Labour
Acronym: OTISMISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Collaborators: Instituto de Saúde Elpidio de Almeida (Unknown); Universidade Federal do Ceara (Other)
Responsible Party: Alex Sandro Rolland de Souza, Instituto de Medicina Integral Prof. Fernando Figueira (IMIP)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORALTIMI
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-10

CONDITIONS: Labor, Induced
Keywords: Misoprostol; Labor, Obstetric; Labor, Induced
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Titrated Misoprostol Solution (Active Comparator)
  Interventions: Drug: Misoprostol
- Vaginal Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Oral solution dose will be 20mcg/hour (misoprostol) or 10ml/hour (placebo) in the first six hours with an increase of 20mcg/hour (10ml/hour) of misoprostol or placebo each six hours if labour does not start, until the maximum dose of 80mcg/hour or 40ml/hour in the first 24 hours.
  Other Names: Prostokos; Cytotec
  Arms: Oral Titrated Misoprostol Solution
Drug: Misoprostol — Vaginal tablets will have 25mcg of misoprostol or placebo.
  Other Names: Prostokos; Cytotec
  Arms: Vaginal Misoprostol

SUMMARY:
The purpose of this study is to compare effectiveness and safety of an oral titrated solution of misoprostol with vaginal misoprostol for induction of labour with an alive fetus.

DETAILED DESCRIPTION:
Several methods for induction of labour are available. However, the most effective and with less frequency of adverse effects is still unknown. Vaginal misoprostol has been used frequently to induce labour but other routes of administrations have been proposed, such as oral, sublingual and, more recently, oral titrated solution. The purpose of this study is to compare effectiveness and safety of this oral misoprostol titrated solution with vaginal misoprostol administration for induction of labour with an alive fetus. A randomized controlled double-blind trial will be carried in three hospitals: Instituto de Medicina Integral Prof. Fernando Figueira, Universidade Federal do Ceará and Instituto de Saúde Elpídio de Almeida, from November 2009 to November 2011. A total of 400 patients must be enrolled. Inclusion criteria are: a) indication for labour induction; b) term pregnancy with alive fetus; Bishop score less than six. Exclusion criteria are: a) age less than 18 years; b) previous uterine scar; c) nonvertex presentation; d) non-reassuring fetal status; e) fetal anomalies; f) fetal growth restriction; g) genital bleeding; h) tumors, malformations and/or ulcers of vulva, perineum or vagina. They will be randomized to receive an oral misoprostol titrated solution with vaginal placebo tablet or oral placebo solution with vaginal misoprostol tablet. Oral solution will have misoprostol at a concentration of 2mcg/ml or placebo. Vaginal tablets will have 25mcg of misoprostol or placebo. Oral solution dose will be 20mcg/hour (misoprostol) or 10ml/hour (placebo) in the first six hours with an increase of 20mcg/hour (10ml/hour) of misoprostol or placebo each six hours if labour does not start, until the maximum dose of 80mcg/hour or 40ml/hour in the first 24 hours. This maximum dose can be maintained for more 24 hours if needed. Vaginal misoprostol or placebo tablets will be administered for each six hours until the maximum dose of 200mcg or eight tablets. Primary outcomes will be vaginal delivery within 24 hours, hyperstimulation syndrome, cesarean section, severe neonatal morbidity or perinatal death, serious maternal morbidity or maternal death. Secondary outcomes will be need of oxytocin for augmentation of labour, number of misoprostol doses needed to bring on labour, interval from first dose to labour and first dose to delivery, failed induction, tachysystole, uterine rupture, need of labour analgesia, instrumental delivery, side effects, maternal death, meconium, non-reassuring fetal heart rate, Apgar scores less than seven at 1st and 5th minutes, admission at neonatal intensive care unit, neonatal encephalopaty, perinatal death and women not satisfied.

ELIGIBILITY:
Inclusion Criteria:

* Indication for labour induction
* Term pregnancy with alive fetus
* Bishop score less than six

Exclusion Criteria:

* Age less than 18 years
* Previous uterine scar
* Nonvertex presentation
* Non-reassuring fetal status
* Fetal anomalies
* Fetal growth restriction
* Genital bleeding
* Tumors, malformations and/or ulcers of vulva, perineum or vagina

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery | 24 hours
Hyperstimulation syndrome | 24 hours
Cesarean section | 3 days
Severe neonatal morbidity or perinatal death | 28 days
Serious maternal morbidity or maternal death | 42

SECONDARY OUTCOMES:
Need of oxytocin for augmentation of labour | 48 hours
Number of doses needed to bring on labour | 48 hours
Interval from 1st dose to labour | 48 hours
Interval from 1st dose to delivery | 48 hours
Failed induction | 72 hours
Tachysystole | 48 hours
Uterine rupture | 72 houras
Need of labour analgesia | 48 hours
Instrumental delivery | 48 hours
Side effects: nausea, vomit, diarrhea, postpartum haemorrhage | 72 hours
Maternal death | 42 days
Meconium | 72 hours
Non-reassuring fetal heart rate | 72 hours
Apgar scores less than 7 at 1st and 5th minute | 1st and 5th minutes after delivery
Admission at neonatal intensive care unit | 28 days
Perinatal or neonatal death | 28 days
Neonatal encephalopathy | 28 days
Women not satisfied with route of drug administration | 48 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Alex SR Souza, Phd student, Study Chair — Professor Fernando Figueira Integral Medicine Institute; Melania MR Amorim, Phd, Study Director — Professor Fernando Figueira Integral Medicine Institute; Aurélio AR Costa, PhD, Principal Investigator — Professor Fernando Figueira Integral Medicine Institute
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira (IMIP), Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Souza AS, Feitosa FE, Costa AA, Pereira AP, Carvalho AS, Paixao RM, Katz L, Amorim MM. Titrated oral misoprostol solution versus vaginal misoprostol for labor induction. Int J Gynaecol Obstet. 2013 Dec;123(3):207-12. doi: 10.1016/j.ijgo.2013.06.028. Epub 2013 Sep 3. PMID 24112746
- [Derived] Orange FA, Passini R Jr, Melo AS, Katz L, Coutinho IC, Amorim MM. Combined spinal-epidural anesthesia and non-pharmacological methods of pain relief during normal childbirth and maternal satisfaction: a randomized clinical trial. Rev Assoc Med Bras (1992). 2012 Jan-Feb;58(1):112-7. PMID 22392325